CLINICAL TRIAL: NCT02336607
Title: A Randomized, Open-label Study to Evaluate the Effects on Blood Pressure Control, Pulse Wave Velocity, as Well as Safety and Tolerability of Felodipine Sustained Release, Alone and in Combination With Metoprolol, Lisinopril or Hydrochlorothiazide, in Chinese Patients With Mild to Moderate Essential Hypertension.
Brief Title: The Effects on Blood Pressure Control, Pulse Wave Velocity, as Well as Safety and Tolerability of Felodipine Sustained Release in Chinese Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: D4385L00001
Record Dates: First submitted 2014-11-25; First posted 2015-01-13 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Felodipine; Single Person; Lisinopril

ARMS (4):
- Felodipine tablet (Plendil) (Experimental)
  Interventions: Drug: Felodipine tablet (Plendil) alone
- Felodipine tablet (Plendil)+Metoprolol tablet (Betaloc ZOK) (Active Comparator)
  Interventions: Drug: Felodipine tablet (Plendil)+Metoprolol tablet (Betaloc ZOK)
- Felodipine tablets (Plendil)+Lisinopril (Zestril) (Active Comparator)
  Interventions: Drug: Felodipine tablets (Plendil)+Lisinopril (Zestril)
- Felodipine tablet (Plendil)+Hydrochlorothiazide (Active Comparator)
  Interventions: Drug: Felodipine tablet (Plendil)+Hydrochlorothiazide

INTERVENTIONS:
Drug: Felodipine tablet (Plendil) alone — Felodipine sustained release tablet single drug therapy (1st week- 2nd week) Eligible subjects will first take felodipine tablet 5mg, once daily, orally for 2 weeks. If blood pressure is controlled after 2 weeks, then the subjects will continue the treatment until the end of primary therapy stage (14th week).
  Arms: Felodipine tablet (Plendil)
Drug: Felodipine tablet (Plendil)+Hydrochlorothiazide — Step 1: Eligible subjects will first take felodipine tablet 5mg, once daily, orally for 2 weeks.
  If blood pressure is not controlled after 2 weeks, then the subjects will go to Step 2: Felodipine sustained release tablet 5mg once daily combined with hydrochlorothiazide 12.5mg, once daily. If blood pressure is not controlled after 4 weeks, then the subjects will go to Step 3: The dosage of felodipine sustained release tablet will be escalated to 10mg, once daily, while the dosage of the combined drug remains the same. If blood pressure is not controlled after 4 weeks, then the subjects will go to Step 4: The dosage of felodipine sustained release tablet keeps 10mg, once daily, while the dosage of different combined drug is doubled.
  Arms: Felodipine tablet (Plendil)+Hydrochlorothiazide
Drug: Felodipine tablet (Plendil)+Metoprolol tablet (Betaloc ZOK) — Step 1: Eligible subjects will first take felodipine tablet 5mg, once daily, orally for 2 weeks.
  If blood pressure is not controlled after 2 weeks, then the subjects will go to Step 2: Felodipine sustained release tablet 5mg once daily combined with metoprolol succinate prolonged-release tablet (Betaloc ZOK) 47.5mg , once daily. If blood pressure is not controlled after 4 weeks, then the subjects will go to Step 3: The dosage of felodipine sustained release tablet will be escalated to 10mg, once daily, while the dosage of the combined drug remains the same. If blood pressure is not controlled after 4 weeks, then the subjects will go to Step 4: The dosage of felodipine sustained release tablet keeps 10mg, once daily, while the dosage of different combined drug is doubled.
  Arms: Felodipine tablet (Plendil)+Metoprolol tablet (Betaloc ZOK)
Drug: Felodipine tablets (Plendil)+Lisinopril (Zestril) — Step 1: Eligible subjects will first take felodipine tablet 5mg, once daily, orally for 2 weeks.
  If blood pressure is not controlled after 2 weeks, then the subjects will go to Step 2: Felodipine sustained release tablet 5mg once daily combined with Lisinopril (Zestril) 10mg, once daily. If blood pressure is not controlled after 4 weeks, then the subjects will go to Step 3: The dosage of felodipine sustained release tablet will be escalated to 10mg, once daily, while the dosage of the combined drug remains the same. If blood pressure is not controlled after 4 weeks, then the subjects will go to Step 4: The dosage of felodipine sustained release tablet keeps 10mg, once daily, while the dosage of different combined drug is doubled.
  Arms: Felodipine tablets (Plendil)+Lisinopril (Zestril)

SUMMARY:
The purpose of this study is to evaluate the effects on blood pressure control, pulse wave velocity, as well as safety and tolerability of felodipine single or combine with other drugs in Chinese Hypertension patients.

DETAILED DESCRIPTION:
In this study, investigators will choose male and female subjects aged between 35 and 79 years old with mild to moderate essential hypertension. At first 2 weeks, all patients will use felodipine 5mg daily. If the blood pressure dosen't meet the target (140/90mmHg), they will be randomized into metoprolol, lisinopril or hydrochlorothiazide combination groups for another 4 weeks therapy. After that, if the blood pressure has still not met the target, up-titrate the felodipine into 10mg, followed by a 4 weeks therapy. And if the blood pressure is still not met the target after that, up-titrate the combine drugs into maximum dosage. The whole treatment duration is 14 weeks.

The primary outcome is to evaluate the percentage of subjects reaching blood pressure target (defined as < 140 / 90 mmHg) after 14 weeks treatment with felodipine sustained release in combination with metoprolol, lisinopril or hydrochlorothiazide.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Female or male aged between 35-79 years old
3. Mild to moderate essential hypertension patients who meet any of the following criterias:

   * Newly diagnosed, drug-naive, or without any antihypertension treatment for at least 3 months, moderate essential hypertension patients. (160mmHg mean SiSBP 180mmHg or 100mmHg mean SiDBP 110mmHg)
   * Newly diagnosed, drug-naive, or without any antihypertension treatment for at least 3 months, mild essential hypertension patients (140mmHg mean SiSBP 160mmHg or 90mmHg mean SiDBP 100mmHg) with high or extreme high cardiovascular risk (a)(having 3 or more than 3 risk factors and/or target organ lesion and/or diabetes mellitus).

     (a) according to Chinese guideline for prevention and treatment of patients with hypertension 2004.
   * The patients have already received starting dosage of single anti-hypertension drug therapy (exclude the drugs containing felodipine component ), however the blood pressure is not well controlled (140mmHg mean SiSBP 160mmHg or 90mmHg mean SiDBP 100mmHg). After stopping the drug for 5 eliminating half life time, the patients meet any one of the following two:

     1. 160mmHg mean SiSBP 180mmHg or 100mmHg mean SiDBP 110mmHg.
     2. 140mmHg mean SiSBP 160mmHg or 90mmHg mean SiDBP 100mmHg) with high or extreme high cardiovascular risk* (having 3 or more than 3 risk factors and/or target organ lesion and/or diabetes mellitus).

Sitting blood pressure is taken after subjects take a seat to rest for 5 minutes before the next medication.

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Known or suspected secondary hypertension
2. Resting heart rate is < 55bpm.
3. Sick sinus syndrome
4. Atrioventricular block of first degree (with P-R>0.24seconds), or second or third degree
5. Other clinical significant arrhythmia
6. Unstable and/or decompensated congestive heart failure
7. Angina, acute myocardial infarction, percutaneous coronary intervention (PCI), or cardiac surgery
8. Asthma or moderate to severe chronic obstructive pulmonary disease
9. Type 1 diabetes mellitus
10. Gout history
11. Fasting serum glucose of greater than 200 mg/dl (11.1 mmol/L) or type 2 diabetes mellitus needs insulin therapy
12. ALT>3ULN
13. Cr>1.5mg/dl
14. Pregnancy or lactation.
15. Alcohol or drug abuse
16. Known need for other concomitant anti-hypertensive therapy during the study besides the study drug.
17. Known or suspected allergy to investigational drug or non-active ingredients of investigational drugs, known allergy to other blockers, calcium antagonist, diuretics, angiotensin converting enzyme inhibitor or with other contraindications.
18. Suspected white-coat hypertension based on investigator's judgement.

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2005-12; Primary Completion 2006-06 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ningling Sun, PhD, MD, Principal Investigator — Beijing University People's Hospital, Department of Cardiology

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=2070&filename=CSR-D4385L00001.pdf
- See also: CSR-D4385L00001.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=2070&filename=CSR-D4385L00001.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled in 10 centers in the People's Republic of China. First patient screened on 26th Dec. 2005, last patient completed last visit on 17th Aug. 2006. A total of 529 patients attended the screening visit. ITT population (481),PP population (390), Safety population (522).
Pre-assignment Details: After enrollment, 7 did not take the test medicine, 522 were given felodipine 5 mg once daily. Of these, 38 patients did not complete the 2-week felodipine monotherapy period.
Groups:
- Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK): Felodipine ER 5mg qd + Metoprolol ER 47.5mg qd; patients who didn't reach the target blood pressure(140/90) after 2 weeks since first administeration,rise dose to Felodipine ER 10mg qd + Metoprolol 47.5mg qd; patients who didn't reach the target blood pressure(140/90) after 2 weeks since first administeration, rise the dose to Felodipine 10mg qd + Metoprolol 95mg qd till the end of the study (week 14).
- Felodipine Tablets (Plendil)+Lisinopril (Zestril): Felodipine ER 5mg qd + Lisinopril 10mg qd; patients who didn't reach the target blood pressure(140/90) after 2 weeks since first administeration,rise dose to Felodipine ER 10mg qd + Lisinopril 10mg qd; patients who didn't reach the target blood pressure(140/90) after 2 weeks since first administeration, rise the dose to Felodipine 10mg qd + Lisinopril 20mg qd till the end of the study ( week 14).
- Felodipine Tablet (Plendil)+Hydrochlorothiazide: Felodipine ER 5mg qd + Hydrochlorothiazide 12.5mg qd; patients who didn't reach the target blood pressure(140/90) after 2 weeks since first administeration,rise dose to Felodipine ER 10mg qd + Hydrochlorothiazide 12.5mg qd; patients who didn't reach the target blood pressure(140/90) after 2 weeks since first administeration, rise the dose to Felodipine 10mg qd + Hydrochlorothiazide 25mg qd till the end of the study (week 14).
- Felodipine Tablet (Plendil): Felodipine ER 5mg qd, the patients who didn't achive the target blood pressure (140/90) after 2 weeks (week1 and week2), switch to combination thearapies.
Period: Overall Study
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Started | 85 | 85 | 92 | 267
Patients Included in ITT Population | 84 | 84 | 91 | 222
Patients Included in PP Population | 78 | 75 | 75 | 162
Patients Included in Safety Population | 85 | 85 | 92 | 260
Completed | 81 | 75 | 86 | 180
Not Completed | 4 | 10 | 6 | 87
Not completed — Physician Decision | 1 | 4 | 3 | 15
Not completed — Lack of Efficacy | 1 | 0 | 0 | 2
Not completed — Lost to Follow-up | 2 | 1 | 0 | 21
Not completed — Protocol Violation | 0 | 1 | 1 | 3
Not completed — Adverse Event | 0 | 2 | 2 | 26
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 20

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are based on ITT group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil) | Total
Number analyzed (Participants) | 84 | 84 | 91 | 222 | 481
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (10.8) | 55.2 (10.7) | 55.6 (9.9) | 55 (11.3) | 54.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 35 | 110 | 215
  Male | 49 | 49 | 56 | 112 | 266

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Reaching Blood Pressure Target (Defined as < 140 / 90 mmHg) After 14 Weeks of Felodipine Sustained Release in Combination With Metoprolol, Lisinopril or Hydrochlorothiazide.
Time Frame: 14 weeks
Population: The ITT population was defined as all patients who received at least one dose of study drug after randomization and had measurements of blood pressure at baseline and from at least one visit after randomization.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Number analyzed (Participants) | 78 | 75 | 75 | 181
Percentage | 74.1 [64.5 to 83.6] | 80.5 [71.7 to 89.4] | 80.2 [71.8 to 88.6] | NA [NA to NA] — Not include in the analysis of primary end point

2. Secondary Outcome: The Percentage of Subjects Reaching Blood Pressure Target (Defined as < 140 / 90 mmHg) After 4 Weeks of Felodipine Sustained Release in Combination With Metoprolol, Lisinopril or Hydrochlorothiazide.
Description: The duration of the combination therapy was 4 weeks. Blood pressure was measured at week 6 of the trial.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Number analyzed (Participants) | 83 | 84 | 91 | 193
Percentage | 45.8 [35.1 to 56.5] | 59.5 [49 to 70] | 46.2 [35.9 to 56.4] | NA [NA to NA] — Not include in the analysis of this end point

3. Secondary Outcome: The Percentage of Subjects Reaching Blood Pressure Target (Defined as < 140 / 90 mmHg) After 8 Weeks of Felodipine Sustained Release in Combination With Metoprolol, Lisinopril or Hydrochlorothiazide.
Description: The duration of the combination therapy was 8 weeks. Blood pressure was measured at week 10 of the trial.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Number analyzed (Participants) | 84 | 81 | 89 | 181
Percentage | 78.6 [69.8 to 87.3] | 79 [70.1 to 87.9] | 78.7 [70.1 to 87.2] | NA [NA to NA] — Not include in the analysis of this end point

4. Secondary Outcome: The Magnitude of Systolic and Diastolic Blood Pressure Change From Baseline Among All Randomized Subjects After 4 Weeks of Felodipine Sustained Release in Combination With Metoprolol, Lisinopril or Hydrochlorothiazide.
Description: The duration of the combination therapy was 4 weeks. Blood pressure was measured at week 6 of the trial.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Number analyzed (Participants) | 83 | 84 | 91 | 193
mmHg
  Change of systolic blood pressure | -10.3 (2.0) | -13.4 (1.8) | -9.8 (1.4) | NA (NA) — Not include in the analysis of this end point
  Change of diastolic blood pressure | -7.3 (1.5) | -9.9 (1.4) | -6.0 (1.0) | NA (NA) — Not include in the analysis of this end point

5. Secondary Outcome: The Magnitude of Systolic and Diastolic Blood Pressure Changes From Baseline Among All Randomized Subjects After 8 Weeks of Felodipine Sustained Release in Combination With Metoprolol, Lisinopril or Hydrochlorothiazide.
Description: The duration of the combination therapy was 8 weeks. Blood pressure was measured at week 10 of the trial.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Number analyzed (Participants) | 84 | 81 | 89 | 181
mmHg
  Change of systolic blood pressure | -17.8 (2.2) | -18.0 (1.9) | -16.4 (1.5) | NA (NA) — Not include in the analysis of this end point
  Change of diastolic blood pressure | -11.3 (1.3) | -12.1 (1.2) | -10.7 (0.9) | NA (NA) — Not include in the analysis of this end point

6. Secondary Outcome: The Magnitude of Systolic and Diastolic Blood Pressure Changes From Baseline Among All Randomized Subjects After 12 Weeks of Felodipine Sustained Release in Combination With Metoprolol, Lisinopril or Hydrochlorothiazide.
Description: The duration of the combination therapy was 12 weeks. Blood pressure was measured at week 14 of the trial.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Number analyzed (Participants) | 81 | 77 | 86 | 181
mmHg
  Change of systolic blood pressure | -16.6 (2.1) | -18.0 (1.9) | -16.8 (1.4) | NA (NA) — Not include in the analysis of this end point
  Change of diastolic blood pressure | -10.7 (1.5) | -12.8 (1.3) | -10.6 (1.0) | NA (NA) — Not include in the analysis of this end point

7. Secondary Outcome: The Magnitude of Systolic and Diastolic Blood Pressure Changes From Baseline Among the Subjects Who Reached Target at 4 Weeks of Felodipine Sustained Release in Combination With Metoprolol, Lisinopril or Hydrochlorothiazide.
Description: The duration of the combination therapy was 4 weeks. Blood pressure was measured at week 6 of the trial.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Number analyzed (Participants) | 38 | 50 | 42 | 190
mmHg
  Change of systolic blood pressure | -16.1 (2.2) | -17.1 (1.6) | -16.4 (1.4) | NA (NA) — Not include in the analysis of this end point
  Change of diastolic blood pressure | -12.3 (1.6) | -10.9 (1.2) | -8.2 (1.0) | NA (NA) — Not include in the analysis of this end point

8. Secondary Outcome: The Magnitude of Systolic and Diastolic Blood Pressure Changes From Baseline Among the Subjects Who Reached Target After 8 Weeks of Felodipine Sustained Release in Combination With Metoprolol, Lisinopril or Hydrochlorothiazide.
Description: The duration of the combination therapy was 8 weeks. Blood pressure was measured at week 10 of the trial.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Number analyzed (Participants) | 66 | 64 | 70 | 180
mmHg
  Change of systolic blood pressure | -19.4 (1.6) | -19.7 (1.4) | -18.5 (1.1) | NA (NA) — Not include in the analysis of this end point
  Change of diastolic blood pressure | -13.4 (1.1) | -13.1 (0.9) | -11.5 (0.7) | NA (NA) — Not include in the analysis of this end point

9. Secondary Outcome: The Magnitude of Systolic and Diastolic Blood Pressure Changes From Baseline Among the Subjects Who Reached Target at 12 Weeks of Felodipine Sustained Release in Combination With Metoprolol, Lisinopril or Hydrochlorothiazide.
Description: The duration of the combination therapy was 12 weeks. Blood pressure was measured at week 14 of the trial.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Number analyzed (Participants) | 60 | 62 | 69 | 176
mmHg
  Change of systolic blood pressure | -18.4 (1.7) | -20.3 (1.5) | -18.2 (1.2) | NA (NA) — Not include in the analysis of this end point
  Change of diastolic blood pressure | -13.0 (1.2) | -13.6 (1.1) | -12.2 (0.8) | NA (NA) — Not include in the analysis of this end point

10. Secondary Outcome: The Change of Pulse Wave Velocity at 12 Weeks Compare With Baseline Data of Felodipine Sustained Release in Combination With Metoprolol, Lisinopril or Hydrochlorothiazide.
Description: The duration of the combination therapy was 12 weeks. The change of pulse wave velocity was measured at week 14 of the trial.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Number analyzed (Participants) | 33 | 32 | 35 | 181
m/s | -0.12 (0.27) | -0.44 (0.38) | -0.06 (0.27) | NA (NA) — Not include in the analysis of this end point

11. Secondary Outcome: The Change of Pulse Wave Velocity From Baseline at 2, 14 Weeks of Felodipine Sustained Release Alone.
Description: as for outcome 10
Time Frame: 12 weeks
Population: The ITT population was defined as all patients who received at least one dose of study drug after randomization and had measurements of The change of pulse wave velocity at baseline and from at least one visit after randomization.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Number analyzed (Participants) | 33 | 32 | 35 | 181
m/s
  week 2 | NA (NA) — Not include in the analysis of this end point | NA (NA) — Not include in the analysis of this end point | NA (NA) — Not include in the analysis of this end point | -0.58 (1.69)
  week 14 | NA (NA) — Not include in the analysis of this end point | NA (NA) — Not include in the analysis of this end point | NA (NA) — Not include in the analysis of this end point | -0.86 (1.93)

12. Secondary Outcome: The Magnitude of Systolic and Diastolic Blood Pressure Changes From Baseline Among the Subjects Who Reached Target at 2 Weeks of Felodipine Sustained Release, Alone
Description: The duration of the combination therapy was 2 weeks. Blood pressure was measured at week 2 of the trial.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Number analyzed (Participants) | 84 | 84 | 91 | 208
mmHg
  Change of systolic blood pressure | NA (NA) — Not include in the analysis of this end point | NA (NA) — Not include in the analysis of this end point | NA (NA) — Not include in the analysis of this end point | -22.8 (11.2)
  Change of diastolic blood pressure | NA (NA) — Not include in the analysis of this end point | NA (NA) — Not include in the analysis of this end point | NA (NA) — Not include in the analysis of this end point | -15.1 (8.2)

ADVERSE EVENTS:
Arm/Group | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) | Felodipine Tablet (Plendil)+Hydrochlorothiazide | Felodipine Tablet (Plendil)
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/85 | 0/92 | 2/260
Other Adverse Events (participants affected / at risk) | 11/85 | 8/85 | 9/92 | 46/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) (N=85) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) (N=85) | Felodipine Tablet (Plendil)+Hydrochlorothiazide (N=92) | Felodipine Tablet (Plendil) (N=260)
Gastrointestinal system damage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — Not considered drug related according to the investigator.
Nervous system damage (Nervous system disorders) | 0 | 0 | 0 | 1 — Not considered drug related according to the investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Felodipine Tablet (Plendil)+Metoprolol Tablet (Betaloc ZOK) (N=85) | Felodipine Tablets (Plendil)+Lisinopril (Zestril) (N=85) | Felodipine Tablet (Plendil)+Hydrochlorothiazide (N=92) | Felodipine Tablet (Plendil) (N=260)
Headache (Nervous system disorders) | 4 | 5 | 4 | 33
Flushing (Vascular disorders) | 7 | 3 | 5 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No